CLINICAL TRIAL: NCT03465306
Title: Developing and Validating Clinical Efficacy for Obesity Digital CBT Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Noom Inc. (Industry); InBody (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: ObesityCBT
Record Dates: First submitted 2018-01-15; First posted 2018-03-14 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-04

CONDITIONS: Search MeSH
Keywords: Obesity; Cognitive Behavioral Therapy
MeSH Terms: conditions — Obesity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This study is been designed to have pre, post, and follow-up phases.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive digital CBT (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Standard digital CBT (Active Comparator)
  Interventions: Device: Self-guided

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive-behavioral therapy is a psycho-social intervention that is the most widely used evidence-based practice for improving mental health and requires active interactions between the participants and a therapist or coach.
  Arms: Intensive digital CBT
Device: Self-guided — Self-guided refers to any contact between the participants and a therapist or coach.
  Arms: Standard digital CBT

SUMMARY:
The aim of the present study is to develop and validate the effects of a new cognitive behavioral therapy (CBT) using digital healthcare mobile apps such as Noom Coach and InBody.

DETAILED DESCRIPTION:
Seventy female participants whose BMI scores were above 23 and who had no other clinical problem except obesity were randomized into an experimental and a control group. Forty-five people in the experimental group were connected with the therapist using digital healthcare apps, so they got daily feedbacks and assignments for 8 weeks. Twenty-five people in the control group also used digital healthcare apps but they were asked to do self-care without intervention.

ELIGIBILITY:
Inclusion Criteria:

* SIMS score ranks over high 20% of total

Exclusion Criteria:

* Had been prescribed with psychological problems or medical problems.

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline | Baseline, at 8 weeks, at 6 months
  Weight difference

SECONDARY OUTCOMES:
weight and height will be combined to report BMI in kg/m^2 | Baseline, at 8 weeks, at 6 months
  BMI difference
Fat percent | Baseline, at 8 weeks, at 6 months
  Fat percent difference
Rosenberg Self-Esteem Scale (RSES). Child / Adolescent Measures | Baseline, at 8 weeks, at 6 months
  Psychological index, total scores range from 10~40, higher the score lower the self-esteem.
Body Shape Questionnaire: Psychometric properties of the short version (BSQ-8C) | Baseline, at 8 weeks, at 6 months
  Psychological index, total scores range from 8~48, higher the score lower the satisfaction to self-body image.
Dutch Eating Behavior Questionnaire (DEBQ) | Baseline, at 8 weeks, at 6 months
  Psychological index, total scores range from 33~165, higher the score more problems in eating behavior.
Yale Food Addiction Scale (YFAS) | Baseline, at 8 weeks, at 6 months
  Psychological index, total scores range from 0~7, higher the score more expected to have food addiction.
Trait Anxiety Inventory (TAI) | Baseline, at 8 weeks, at 6 months
  Psychological index, total scores range from 20~80, higher the score higher in feelings of anxiety.
Korean Beck Depression Inventory (K-BDI) | Baseline, at 8 weeks, at 6 months
  Psychological index, total scores range from 0~63, higher the score higher in feelings of depressed.
Automatic Thoughts Questionnaire-30 (ATQ-30) | Baseline, at 8 weeks, at 6 months
  Psychological index, total scores range from 30~150, higher the score higher tendency to have negative automatic thoughts.
the result of cholesterol total | Baseline, at 8 weeks
  Biological index
the result of triglycerides (TG) | Baseline, at 8 weeks
  Biological index
the result of gamma-glutamyl transferase (GGT) | Baseline, at 8 weeks
  Biological index
the result of glucose | Baseline, at 8 weeks
  Biological index
the result of alanine aminotransferase (ALT) | Baseline, at 8 weeks
  Biological index
the result of aspartate aminotransferase (AST) | Baseline, at 8 weeks
  Biological index
the result of insulin | Baseline, at 8 weeks
  Biological index
the result of leptin | Baseline, at 8 weeks
  Biological index
Buffet index | Baseline, at 8 weeks
  Buffet test, total scores range from 0~100, higher the score better in healthy food choice and amount of intake.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882
- [Derived] Kim M, Lee S, Cho E, Hong KW, You SJ, Choi HJ. CETP and APOA2 polymorphisms are associated with weight loss and healthy eating behavior changes in response to digital lifestyle modifications. Sci Rep. 2023 Dec 7;13(1):21615. doi: 10.1038/s41598-023-48823-w. PMID 38062157
- [Derived] Kim M, Yang J, Ahn WY, Choi HJ. Machine Learning Analysis to Identify Digital Behavioral Phenotypes for Engagement and Health Outcome Efficacy of an mHealth Intervention for Obesity: Randomized Controlled Trial. J Med Internet Res. 2021 Jun 24;23(6):e27218. doi: 10.2196/27218. PMID 34184991
- [Derived] Kim M, Kim Y, Go Y, Lee S, Na M, Lee Y, Choi S, Choi HJ. Multidimensional Cognitive Behavioral Therapy for Obesity Applied by Psychologists Using a Digital Platform: Open-Label Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Apr 30;8(4):e14817. doi: 10.2196/14817. PMID 32352391